CLINICAL TRIAL: NCT02937922
Title: Effect of Aerobic Exercise, Resistance or Combined in Endothelial Injury in Hypertensive Patients
Brief Title: Effect of Exercise on Endothelial Injury in Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Gustavo Waclawovsky, Principal Investigator, Instituto de Cardiologia do Rio Grande do Sul
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: Endothelial
Record Dates: First submitted 2016-10-14; First posted 2016-10-19 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Hypertension; Healthy
Keywords: Exercise; Endothelium; Hypertension; Endothelial progenitor cell; Endothelial microparticle
MeSH Terms: conditions — Hypertension; Motor Activity | interventions — Exercise; Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AEROBIC (Active Comparator): The aerobic exercise session (AE) will consist of 40 minutes on an exercise bike in heart rate (HR) corresponding to 60% of heart rate reserve (moderate intensity) acquired by the formula of Karvonen: [(HR max - HR rest) x desired intensity] + HR rest; monitored through heart monitor brand Polar and perceived exertion rating (Borg scale of 6-20). It will be added to the exercise time 5-7 minutes to proper heating.
  Interventions: Other: AEROBIC
- RESISTANCE (Active Comparator): The resistance exercise session (RE) will last 40 minutes and will consist in carrying out 4 sets of 12 repetitions with interval of 90 seconds between sets and exercises. The weight will be adjusted to 60% of a maximum repetition (1-RM) in four exercise for the lower limbs: leg press, knee extension, bend knees and plantar flexion (calf). The cadence of each series will be controlled by electronic metronome and performed with 2 seconds in the concentric phase and 2 seconds in the eccentric phase. It will be added to the exercise time 5-7 minutes for the warming to be held in the leg press exercise (one set of 15 to 20 repetitions with 1/3 load set for the session).
  Interventions: Other: RESISTANCE
- COMBINED (Active Comparator): The combined exercise session (resistance and aerobic) will last 40 minutes. The exercise resistance phase of the combined session will consist of 20 minutes, according to the resistance exercise described above. Immediately after resistance exercise, patients will perform aerobic exercise (AE) for 20 minutes. In order to keep the equivalent time among the three interventions (aerobic exercise resistance and combined) will be performed two series (2 x 12 repetitions) in each resistance exercise.
  Interventions: Other: COMBINED

INTERVENTIONS:
Other: AEROBIC — The aerobic exercise session (AE) will consist of 40 minutes on an exercise bike in heart rate (HR) corresponding to 60% of heart rate reserve (moderate intensity) acquired by the formula of Karvonen: [(HR max - HR rest) x desired intensity] + HR rest; monitored through heart monitor brand Polar and perceived exertion rating (Borg scale of 6-20). It will be added to the exercise time 5-7 minutes to proper heating.
  Other Names: Aerobic exercise
  Arms: AEROBIC
Other: RESISTANCE — The resistance exercise session (RE) will last 40 minutes and will consist in carrying out 4 sets of 12 repetitions with interval of 90 seconds between sets and exercises. The weight will be adjusted to 60 % of a maximum repetition (1-RM) (moderate intensity) in four exercise for the lower limbs: leg press, knee extension, bend knees and plantar flexion (calf). The cadence of each series will be controlled by electronic metronome and performed with 2 seconds in the concentric phase and 2 seconds in the eccentric phase. It will be added to the exercise time 5-7 minutes for the warming to be held in the leg press exercise (one set of 15 to 20 repetitions with 1/3 load set for the session).
  Other Names: Resistance exercise
  Arms: RESISTANCE
Other: COMBINED — The combined exercise session (resistance and aerobic) will last 40 minutes. The exercise resistance phase of the combined session will consist of 20 minutes, according to the resistance exercise described above. Immediately after resistance exercise, patients will perform aerobic exercise (AE) for 20 minutes. In order to keep the equivalent time among the three interventions (aerobic exercise, resistance and combined) will be performed two series (2 x 12 repetitions) in each resistance exercise.
  Other Names: Combined exercise
  Arms: COMBINED

SUMMARY:
Introduction: Endothelial dysfunction precedes atherosclerosis being evidenced in patients with hypertension. Increasing physical activity levels and/or physical exercise are part of the recommendations of antihypertensive therapy. However, the effects of oscillations and/or increase the systemic blood pressure induced by exercise session on endothelial function has not been studied.

Objective: To evaluate the effect of aerobic exercise, resistance exercise and combined exercise on endothelial injury levels in patients with hypertension.

Methodology: Hypertensive (n = 51) and healthy subjects (n = 30) (30-59 years old) will perform at random 40 minutes of aerobic exercise (50-60% of heart rate reserve) or 40 minutes of resistance exercise (4 x 12 repetitions of exercises for lower limbs, 60-70% of one repetition maximum and 60-90 second interval) or 40 minutes of combined exercise (20 minutes of resistance exercise and 20 minutes of aerobic exercise, in that order). Blood will be collected 10 minutes before, 10 and 60 minutes after intervention for the quantification of endothelial microparticles (MPE) circulating (induced endothelial lesion) and endothelial progenitor cells (EPC) circulating (endothelial recovery capacity) by flow cytometry. Ambulatory blood pressure monitoring (ABPM) will be held before and after the intervention. Ultrasonography is used to measure the flow-mediated dilation of the brachial artery 10 minutes before, 10, 30 and 60 minutes after the intervention.

Statistics: generalized estimating equation (GEE) for repeated measurements and Person correlation, being significant p < 0.05.

It is expected to show results to ensure cardiovascular protection in patients with hypertension caused by different types of exercise and consequent endothelial injury and release induced regenerative factors. Knowledge of the magnitude of injury and endothelial recovery provided by different types of exercise can contribute scientifically to health professionals aimed at prescribing exercise with a vascular protective vision in patients with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Adults with hypertension;
* 30 to 59 years old.

Exclusion Criteria:

* Diabetes;
* Heart disease;
* Participating in any regular exercise program over the last six months;
* Orthopedic impairments or any physical or mental limitation that prevents - achievement of physical exercise;
* Body Mass Index in class II obesity or more (BMI ≥ 35 kg / m2);
* Smoking.

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2016-01; Primary Completion 2019-12 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Effects of exercise on the percentage of circulating endothelial progenitor cells analyzed by flow cytometry in patients with hypertension | two years

SECONDARY OUTCOMES:
Effects of exercise on the number of circulating endothelial microparticles analyzed by flow cytometry in patients with hypertension | two years

IPD SHARING:
Plan to Share IPD: Yes
Data will be presented to participants from lectures.

REFERENCES:
- [Background] Waclawovsky G, Umpierre D, Figueira FR, De Lima ES, Alegretti AP, Schneider L, Matte US, Rodrigues TC, Schaan BD. Exercise on Progenitor Cells in Healthy Subjects and Patients with Type 1 Diabetes. Med Sci Sports Exerc. 2016 Feb;48(2):190-9. doi: 10.1249/MSS.0000000000000764. PMID 26312614
- [Background] Amabile N, Cheng S, Renard JM, Larson MG, Ghorbani A, McCabe E, Griffin G, Guerin C, Ho JE, Shaw SY, Cohen KS, Vasan RS, Tedgui A, Boulanger CM, Wang TJ. Association of circulating endothelial microparticles with cardiometabolic risk factors in the Framingham Heart Study. Eur Heart J. 2014 Nov 7;35(42):2972-9. doi: 10.1093/eurheartj/ehu153. Epub 2014 Apr 16. PMID 24742886